CLINICAL TRIAL: NCT06767462
Title: A Multicentre Study Assessing Ophthalmic Safety in Patients With Breast Cancer
Brief Title: An Ophthalmic Safety Study in Patients With Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D853AC00001
Record Dates: First submitted 2024-11-15; First posted 2025-01-10 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Ophthalmic Safety in Patients With Breast Cancer
Keywords: Ophthalmic Safety assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — No human sample collection in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1 from Qualifying Study
- Cohort 2 from Qualifying Study

SUMMARY:
To assess ophthalmic health in parallel cohorts of patients with breast cancer

DETAILED DESCRIPTION:
This is a multicentre study assessing the ophthalmic safety in patients who are participating in a qualifying study. The study will include two cohorts of at least 60 individuals each.

To be able to account for events associated with aging, worsening of pre-existing conditions, etc., ophthalmic study assessments will be performed in parallel in two cohorts at the same timepoints. The duration of the study assessment period will be approximately 12 months. Longer duration of the study would result in additional patient burden.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent in the qualifying study.
2. Signed informed consent in the ophthalmic study prior to any ophthalmic study specific assessments and procedures.
3. Completed the baseline ophthalmic examination for this study before the first dose in the qualifying study.
4. Meets all the eligibility criteria in the qualifying study

Exclusion Criteria:

1. Patients not randomized and not receiving study assigned treatment in a qualifying study.
2. Patients with contraindications to any ophthalmic procedure required by the study or sensitivity/allergy to pupil dilating agents.
3. Judgement by the investigator that the patient should not participate in the ophthalmic study if the patient is unlikely to comply with study procedures, restrictions, and requirements

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are currently participating in qualifying studies
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2027-07-06 (Estimated); Study Completion 2027-07-06 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity Testing (Snellen units) | Ophthalmic review by central reader until 28 days after End of Study visit.
  To detect potential impairment in central vision in patients with breast cancer.
Slit Lamp examination (normal/abnormal) | Ophthalmic review by local ophthalmologist until 28 days after End of Study visit.
  To detect any corneal changes or lens changes (eg, cataracts) that could impact high and low contrast acuity/visual field in patients with breast cancer.
Optical Coherence Tonometry (μm) | Ophthalmic review by central reader until 28 days after End of Study visit.
  To assess any structural change/damage to the eye or any long-term visual effects in patients with breast cancer.
Fundus Examination (normal/abnormal) | Ophthalmic review by central reader until 28 days after End of Study visit.
  To assess any structural change/damage to the eye or any long-term visual effects in patients with breast cancer.

SECONDARY OUTCOMES:
Incidence and Severity of Adverse Events, with Severity Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI-CTCAE v5.0) | Until 28 days after the End of Study visit
  To assess the ophthalmic safety in patients with breast cancer.

CONTACTS AND LOCATIONS:
Locations (61):
- United States (12):
  - Research Site, La Jolla, California
  - Research Site, Palo Alto, California
  - Research Site, San Diego, California
  - Research Site, Iowa City, Iowa
  - Research Site, New York, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Clairton, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Bartlett, Tennessee
  - Research Site, Houston, Texas
- Argentina (4):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Córdoba
  - Research Site, San Miguel de Tucumán
- Belgium (3):
  - Research Site, Edegem
  - Research Site, Leuven
  - Research Site, Liège
- Brazil (11):
  - Research Site, Alfenas
  - Research Site, Belo Horizonte
  - Research Site, Curitiba
  - Research Site, Lajeado
  - Research Site, Porto Alegre
  - Research Site, Pouso Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
  - Research Site, Sorocaba
  - Research Site, Três Lagoas
  - Research Site, Vitória
- Research Site, Montreal, Quebec, Canada
- Research Site, Santiago, Chile
- France (5):
  - Research Site, Bordeaux Cédex
  - Research Site, Caen
  - Research Site, Nantes
  - Research Site, Poitiers
  - Research Site, Suresnes
- Israel (2):
  - Research Site, Ashdod
  - Research Site, Nahariya
- Research Site, Milan, Italy
- Mexico (4):
  - Research Site, Aguascalientes
  - Research Site, Mexico City
  - Research Site, San Pedro Garza García
  - Research Site, Veracruz
- Poland (2):
  - Research Site, Lodz
  - Research Site, Nowa Sól
- Portugal (3):
  - Research Site, Amadora
  - Research Site, Braga
  - Research Site, Lisbon
- South Korea (3):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Seoul
- Spain (9):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Girona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Leganés
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Salamanca
  - Research Site, Sant Joan Despí

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: http://www.vivli.org/